CLINICAL TRIAL: NCT02266888
Title: B Cell Targeted Induction to Improve Outcomes in Pediatric Lung Transplantation (CTOTC-08)
Brief Title: B Cell Induction in Pediatric Lung Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation in Children (Other); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT CTOTC-08; NIAID CRMS ID#: 20181 (Other: DAIT NIAID)
Record Dates: First submitted 2014-10-08; First posted 2014-10-17 (Estimated); Results first posted 2020-07-16 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Lung Transplant
Keywords: B cells; lung transplant recipient; rituximab; placebo; standard of care
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab Induction (Experimental): Rituximab (Rituxan®) Induction Therapy Plus Standard of Care Immunosuppression (thymoglobulin induction, tacrolimus or equivalent, mycophenolate mofetil (MMF) or equivalent, and steroids)
  Interventions: Biological: Rituximab (Rituxan®)
- Placebo Induction (Placebo Comparator): Placebo Induction Therapy Plus Standard of Care Immunosuppression (Thymoglobulin® induction, tacrolimus or equivalent, mycophenolate mofetil (MMF) or equivalent, and steroids)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Rituximab (Rituxan®) — 2 Doses: 375 mg/m^2 on Day 0 (within 12 hours of return to ICU following transplant) and Day 12 (+/-2 days).
  Other Names: Rituxan®
  Arms: Rituximab Induction
Biological: Placebo — Placebo for Rituximab (Rituxan®). 2 Doses: 375 mg/m^2 on Day 0 (within 12 hours of return to ICU following transplant) and Day 12 (+/-2 days).
  Arms: Placebo Induction

SUMMARY:
In this study, doctors are trying to see if a study drug called rituximab (Rituxan®) will lower the number of B cells in the body. Doctors are also trying to see if decreasing B cells with rituximab (Rituxan®) can prevent injury to the transplanted lung. This treatment has been studied in other types of solid organ transplants.

DETAILED DESCRIPTION:
Patients who receive a lung transplant are at risk for rejection of the transplanted lung(s). Rejection occurs when the new lung triggers the body's defense (immune) system. When the immune system is triggered special cells are sent out to destroy the new lung and eventually the lung may not be able to function as it should. These special cells include B cells. B cells are an important part of the immune system and help the body fight infection. One way B cells fight infection is by producing antibodies. B cells and the antibodies they produce are involved in some kinds of rejection after organ transplantation.

ELIGIBILITY:
Inclusion Criteria:

Enrollment:

1. Subject and/or parent guardian must be able to understand and provide informed consent;
2. Candidate for a primary lung transplant (listed for lung transplant);
3. Female and male subjects with reproductive potential must agree to use FDA approved methods of birth control for 12-months after completion of treatment.
4. Adequate bone marrow functions based on the following criteria:

   * Absolute neutrophil count (ANC): >1000mm^3
   * Platelets: >100,000/mm^3
   * Hemoglobin: >7 gm/dL
   * AST or ALT< 2x Upper Limit of Normal unless related to primary disease

Randomization:

Individuals who meet all of the following criteria are eligible for randomization:

1. Serum IgG immunoglobulin level greater than lower level of normal for age based on local laboratory ranges or 400mg/dL within 90 days prior to randomization;
2. Female subjects of childbearing potential must have a negative pregnancy test within 4 hours of transplant;
3. Negative for Hepatitis B infection (if at time of transplant, participant does not exhibit effective immunization, the participant should be re-tested).

Exclusion Criteria:

Enrollment:

Individuals who meet any of these criteria are not eligible for enrollment as study participants:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol;
2. Multi-organ transplant;
3. Previous treatment with rituximab (Rituxan®);
4. History of severe allergic anaphylactic reactions to humanized or murine monoclonal antibodies;
5. History of severe reaction to previous therapy with intravenous immunoglobulin (IVIG);
6. History of Burkholderia cenocepacia;
7. History of anti-CD20 therapy;
8. Persistent hypogammaglobulinemia (IgG < lower level of normal for age based on local laboratory ranges or 400 gm/dL for >2 months) and/or IVIG replacement therapy;
9. Positive blood culture, sepsis or other disease process with hemodynamic instability at time of enrollment;
10. Any history of serologic positivity to HIV, HBsAg, HBcAb and HCV Ab;
11. History of malignancy less than 2 years in remission of malignancy (any history of adequately treated in-situ cervical carcinoma, or adequately treated basal or squamous cell carcinoma of the skin will be permitted);
12. Any condition, including psychiatric disorders, that in the opinion of the investigator would interfere with the subject's ability to comply with study requirements;
13. Participation in another investigational trial within 4 weeks of enrollment;
14. Currently lactating or plans to become pregnant during the timeframe of the study follow-up period;
15. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Randomization:

Individuals who meet any of these criteria are not eligible for randomization:

1. Use of an induction agent other than Thymoglobulin®;
2. Renal insufficiency requiring hemodialysis or ultrafiltration;
3. Inability to obtain intravenous access;
4. Positive blood culture, sepsis or other disease process with hemodynamic instability at time of transplant;
5. Use of investigational agent(s) within 5 half-lives of the investigational drug or 4 weeks, whichever is longer;
6. Receipt of a MMR vaccine within 30 days prior to randomization;
7. Any condition that, in the opinion of the investigator, would interfere with the subject's ability to comply with study requirements.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Sweet, M.D., Ph.D., Study Chair — Washington University Medical Center: Department of Pediatrics, Division of Allergy, Immunology and Pulmonary Medicine; Lara Danziger-Isakov, M.D., M.P.H., Study Chair — Cincinnati Children's Hospital: Division of Infectious Diseases
Locations (7):
- United States (7):
  - Stanford University, Palo Alto, California
  - Children's Hospital Boston, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- [Result] Sweet SC, Armstrong B, Blatter J, Chin H, Conrad C, Goldfarb S, Hayes D Jr, Heeger PS, Lyou V, Melicoff-Portillo E, Mohanakumar T, Odim J, Ravichandran R, Schecter M, Storch GA, Visner G, Williams NM, Danziger-Isakov L. CTOTC-08: A multicenter randomized controlled trial of rituximab induction to reduce antibody development and improve outcomes in pediatric lung transplant recipients. Am J Transplant. 2022 Jan;22(1):230-244. doi: 10.1111/ajt.16862. Epub 2021 Nov 5. PMID 34599540
- [Result] Duncan-Park S, Dunphy C, Becker J, D'Urso C, Annunziato R, Blatter J, Conrad C, Goldfarb SB, Hayes D Jr, Melicoff E, Schecter M, Visner G, Armstrong B, Chin H, Kesler K, Williams NM, Odim JN, Sweet SC, Danziger-Isakov L, Shemesh E. Remote intervention engagement and outcomes in the Clinical Trials in Organ Transplantation in Children consortium multisite trial. Am J Transplant. 2021 Sep;21(9):3112-3122. doi: 10.1111/ajt.16567. Epub 2021 Apr 12. PMID 33752251
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Clinical Trials in Organ Transplantation in Children (CTOT-C) — http://www.ctotc.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven sites in the United States enrolled 45 participants into this trial.
Groups:
- Rituximab: Induction: Rituximab was administered in two 375 mg/m^2 doses: on Day 0 within 12 hours of return to ICU following transplant and on Day 12 (+/-2 days). Standard of care immunosuppression (thymoglobulin induction, tacrolimus or equivalent, MMF or equivalent, and steroids) was also utilized at each site.
- Placebo: Induction: Rituximab placebo was administered in two 375 mg/m^2 doses: on Day 0 within 12 hours of return to ICU following transplant and on Day 12 (+/-2 days). Standard of care immunosuppression (thymoglobulin induction, tacrolimus or equivalent, MMF or equivalent, and steroids) was also utilized at each site.
- Discontinued Pre-Transplant: Participants who enrolled, but withdrew from the study prior to receiving a transplant.
- Discontinued Pre-Randomization: Participants who were enrolled and transplanted on study, but withdrew from the study prior to randomization.
Period: Overall Study
Arm/Group | Rituximab | Placebo | Discontinued Pre-Transplant | Discontinued Pre-Randomization
Started | 15 | 12 | 11 | 7
Completed | 8 | 8 | 0 | 0
Not Completed | 7 | 4 | 11 | 7
Not completed — Death | 2 | 2 | 4 | 2
Not completed — Physician Decision | 0 | 1 | 2 | 2
Not completed — Study Terminated | 5 | 1 | 0 | 0
Not completed — No Longer Eligible | 0 | 0 | 0 | 2
Not completed — Randomization Closed | 0 | 0 | 4 | 0
Not completed — Personnel unavailable at transplant | 0 | 0 | 0 | 1
Not completed — Transfer of care | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population, defined as all randomized participants who receive at least a portion of the initial rituximab or placebo infusion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab | Placebo | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 11 | 26
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.5 (4.55) | 13.2 (4.47) | 12.8 (4.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 10 | 8 | 18
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 12 | 10 | 22
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 12 | 27
Pre-Transplant Lung Allocation Score (LAS) Diagnosis Group [Count of Participants; unit: Participants] — The Lung Allocation Score (LAS) diagnosis group characterizes a person's lung disease into one of four groups: A, B, C, or D. Group A includes obstructive lung diseases like emphysema and chronic obstructive pulmonary disease. Group B includes pulmonary vascular diseases like hypertension. Group C includes cystic fibrosis and bronchiectasis. Group D includes restrictive diseases like pulmonary fibrosis.
  Participants
    Group A | 1 | 0 | 1
    Group B | 1 | 0 | 1
    Group C | 8 | 10 | 18
    Group D | 5 | 2 | 7
Donor and Recipient Gender [Count of Participants; unit: Participants] — This measure summarizes the cross-tabulation of donor and recipient gender (e.g., Female Donor and Male Recipient).
  Participants
    Female Donor, Female Recipient | 5 | 3 | 8
    Female Donor, Male Recipient | 1 | 0 | 1
    Male Donor, Female Recipient | 3 | 3 | 6
    Male Donor, Male Recipient | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Earliest Time to Any of the Following Events: Chronic Allograft Dysfunction, Listed for Retransplant or Death
Description: This composite outcome measures is defined as the earliest time post-transplant to any of the following events during the follow-up period:
  * Chronic Allograft Dysfunction (defined as the occurrence of confirmed Bronchiolitis Obliterans Syndrome (BOS) grade 0-p or higher or a diagnosis of Obliterative Bronchiolitis (OB)),
  * Listed for re-transplant (e.g., second lung transplant), or
  * Death.
Time Frame: Up to 35 months post-transplant
Population: Intent-to-treat population included all randomized participants who received at least a portion of the initial rituximab or placebo infusion.
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 15 | 12
Days | NA [NA to NA] — The median time to event was not reached due to insufficient number of events. Data is not estimable. | 703 [306 to NA] — The upper confidence limit is not estimable since no events occurred after reaching median survival.
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Test type: Superiority; p = 0.514, Regression, Cox; Hazard Ratio (HR) = 0.673, 90% CI 2-sided [0.248 to 1.826] — Hazard ratio estimated for Rituximab vs. Placebo

2. Secondary Outcome: Percent of Participants Diagnosed With Chronic Allograft Dysfunction
Description: Chronic allograft dysfunction is defined as Bronchiolitis Obliterans Syndrome (BOS) ≥Grade 0p according to the International Society for Heart and Lung Transplantation (ISHLT) criteria, or biopsy proven histologic evidence of obliterans bronchiolitis.
  BOS is an indicator of post-transplant loss of lung function, a sign of allograft dysfunction that presents as a persistent decline in forced expiratory volume in 1 second (FEV1) or forced expiratory flow (FEF) 25-75% (often accompanied by evidence of airway obstruction) that is not the result of other causes such as acute rejection, acute infection, and/or airway stenosis.
  * BOS grade: Spirometry % of baseline
  * 0: FEV1 >90% and FEF25-75% >75%
  * 0-p: FEV1 81-90% and FEF25-75% ≤75%
  * 1: FEV1 66-80%
  * 2: FEV1 51-65%
  * 3: FEV1 ≤50%
Time Frame: Up to 35 months post-transplant
Population: Intent-to-treat population included all randomized participants who 1.) Received at least a portion of the initial rituximab or placebo infusion and 2.) Had at least one biopsy evaluable for OB and sufficient pulmonary function tests for evaluation of BOS.
Measure: Number (90% Confidence Interval); unit: Percent of Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 14 | 11
Percent of Participants | 28.6 [8.7 to 48.4] | 27.3 [5.2 to 49.4]

3. Secondary Outcome: Percent of Participants Listed for Re-Transplant During the Study Follow-Up Period
Description: Participants with a reported date of listing for a second lung transplant during the study follow-up period.
Time Frame: Up to 35 months post-transplant
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percent of Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 15 | 12
Percent of Participants | 0 [0 to 0] | 8.3 [0 to 21.5]

4. Secondary Outcome: Percent of Participants Who Died During the Study Follow-Up Period
Description: Participants with a reported date of death were considered to have met this outcome.
Time Frame: Up to 35 months post-transplant
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percent of Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 15 | 12
Percent of Participants | 13.3 [0 to 27.8] | 25.0 [4.4 to 45.6]

5. Secondary Outcome: Percent of Participants With Primary Graft Dysfunction (PGD)
Description: The International Society for Heart and Lung Transplantation's (ISHLT) grading for Primary Graft Dysfunction (PGD) was used. The severity of PGD is graded 0 - 3 based on the presence or absence of diffuse opacities on chest radiograph and the ratio of arterial oxygen pressure to inspired oxygen concentration. The grading system predicts post-lung transplant outcomes with Grade 3 being the worse.
  Participants were classified as having PGD if graded as 2 or 3 at any time during the first 72 hours post-transplant.
Time Frame: Up to 72 hours post-transplant
Population: Intent-to-treat population included all randomized participants who received at least a portion of the initial rituximab or placebo infusion and had available blood gas (e.g., arterial oxygen pressure) data during the first 72 hours post-transplant.
Measure: Number (90% Confidence Interval); unit: Percent of Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 12 | 7
Percent of Participants | 25.0 [4.4 to 45.6] | 14.3 [0 to 36.0]
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Test type: Superiority; p > 0.999, Fisher Exact

6. Secondary Outcome: Percent of Participants With Occurrence of Grade A Acute Rejection
Description: Pulmonary allograft rejection was defined according to the 2007 International Society for Heart and Lung Transplantation's (ISHLT). Each transbronchial biopsy (TBBx) was evaluated by the local center's pathologist and graded as described below.
  Acute Cellular Rejection (ACR) Grade Classification:
  * A0: None
  * A1: Minimal
  * A2: Mild
  * A3: Moderate
  * A4: Severe
  Participants met this outcome if at any point in time their biopsy was classified as A2, A3, or A4.
Time Frame: Up to 24 months post-transplant
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percent of Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 15 | 12
Percent of Participants | 13.3 [0 to 27.8] | 16.7 [0 to 34.4]
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Test type: Superiority; p > 0.999, Fisher Exact

7. Secondary Outcome: Percent of Participants With Occurrence of Antibody Mediated Rejection
Description: Antibody Mediated Rejection (AMR) was defined based on the revision of the 1996 Working Formulation for the Standardization of Nomenclature in the Diagnosis of Lung Rejection, the Pathology of pulmonary AMR and the 2012 update from the Pathology Council of the International Society for Heart and Lung Transplantation (ISHLT).
  AMR was diagnosed locally and graded as:
  * Grade I: Latent humoral response - Donor Specific Antibody (DSA) or autoantibody present and absence of both abnormal histology and unexplained graft dysfunction
  * Grade II: Subclinical humoral rejection - DSA or autoantibody present and abnormal histology present with an absence of unexplained graft dysfunction
  * Grade III: Humoral rejection - DSA or autoantibody present and abnormal histology present and unexplained graft dysfunction present.
  Higher grades indicate more severe AMR.
  Participants were considered to have met this outcome if at any point in time their biopsy was classified as Grade II or III.
Time Frame: Up to 24 months post-transplant
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percent of Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 15 | 12
Percent of Participants | 0 [0 to 0] | 16.7 [0 to 34.4]
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Test type: Superiority; p = 0.188, Fisher Exact

8. Secondary Outcome: Percent of Participants Meeting Tacrolimus Variability Threshold
Description: Tacrolimus trough levels are generally collected post-transplant to allow clinicians to monitor transplant recipients' adherence to prescribed tacrolimus dosing. This outcome was designed for research purposes as an indicator of adherence to tacrolimus over time.
  Beginning at 3 months post-transplant, a rolling standard deviation (SD) was estimated for each participant who had at least 3 outpatient trough levels collected and recorded. The estimated SD could derive from up to 1 year worth of trough levels at any given time. The larger the SD (variation) of tacrolimus levels, the greater the nonadherence of participant(s) taking tacrolimus as prescribed. Nonadherence is a major reason for post-transplant morbidity.
  Participants were considered to have met this outcome, the tacrolimus variability threshold, if their estimated SD of tacrolimus medication levels at any time was 2.0 ng/mL or greater.
Time Frame: Up to 24 months post-transplant
Population: Intent-to-treat population included all randomized participants who received at least a portion of the initial rituximab or placebo infusion and who had at least 3 outpatient tacrolimus trough levels collected that were at least 3 months post-transplant.
Measure: Number (90% Confidence Interval); unit: Percent of Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 15 | 11
Percent of Participants | 93.3 [82.7 to 100] | 100 [100 to 100]

9. Secondary Outcome: Percent of Participants Meeting Tacrolimus Variability Threshold Who Completed Tacrolimus Variability Intervention
Description: For participants who met the Tacrolimus Variability Threshold and agreed to participate in the Tacrolimus Variability Intervention (TVI), a series of calls with the participant, parent(s)/guardian(s), and trained call center personnel were conducted to address barriers to adherence.
  Refer to Outcome Measure 8 for a description of tacrolimus variability threshold methodology.
Time Frame: Up to 27 months post-transplant
Population: Intent-to-treat population included all randomized participants who received at least a portion of the initial rituximab or placebo infusion, which was subset to participants who qualified for and agreed to participate in the TVI.
Measure: Number (90% Confidence Interval); unit: Percent of Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 7 | 8
Percent of Participants | 85.7 [64.0 to 100] | 100 [100 to 100]

10. Secondary Outcome: Magnitude of Change in Standard Deviation of Tacrolimus Levels Following Intervention
Description: Standard deviation (SD) is a number that describes how a group of measurements are spread out around the average value for that group. A low SD value means the numbers are close to the average; a high SD means the numbers are more spread out. The change in SD of tacrolimus levels was calculated by subtracting each participant's pre-intervention SD from their SD 180 days after enrollment into the intervention (i.e., value of SD 180 days after enrollment minus value of SD before enrollment). A change less than zero (i.e., a negative number) would indicate a decrease in SD, which is good, possibly as a result of the intervention.
Time Frame: Up to 19 months post-transplant
Population: Intent-to-treat population included all randomized participants who received at least a portion of the initial rituximab or placebo infusion, which was subset to participants who qualified for and agreed to participate in the TVI and who had both a pre-TVI and post-TVI measurement available.
Measure: Mean (Standard Deviation); unit: Standard deviation per participant
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 7 | 7
Standard deviation per participant
  Pre-TVI enrollment | 3.95 (1.664) | 5.18 (2.423)
  180 Days after TVI enrollment | 3.03 (0.948) | 2.86 (1.636)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; This is not a comparison between treatment groups, but rather a comparison between timepoints.The Rituximab and Placebo groups were combined for purposes of testing the hypothesis that there would be no change in SD between pre-enrollment and 180 days post-enrollment into the TVI; Test type: Superiority; p = 0.015, Paired t-Test; Mean Difference (Net) = -1.62, 90% CI 2-sided [-2.64 to -0.60]

11. Secondary Outcome: Percent of Participants Experiencing an Infection Episode
Description: Defined by:
  * A local report of bacterial, fungal, or viral infection through either the organism specific case report form (CRF) or adverse event reporting; or
  * Presence of symptoms at the time of a study visit without a local report of infection but with a corresponding Core Lab identified viral infection
    * All symptoms reported at the time of a study visit were evaluated for any Epstein-Barr Virus (EBV) and Cytomegalovirus (CMV) infections identified by the Core Lab
    * For any other infections identified in Core Lab Nasopharyngeal (NP) and Bronchoalveolar Lavage (BAL) biospecimens: shortness of breath, new x-ray or other imaging finding, new supplemental oxygen requirement, cough with sputum, and decreased spirometry were evaluated signs/symptoms.
  Participants were considered to have met this outcome if at any point in time they had an infection meeting the referenced criteria.
Time Frame: Up to 24 months post-transplant
Population: as for outcome 1
Measure: Number; unit: Percent of Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 15 | 12
Percent of Participants | 100 | 100

12. Secondary Outcome: Number of Participants With Severity of Infection Episodes
Description: The severity of infection episodes was determined by the site Principal Investigator (PI) using the adverse event (AE) scale of mild to moderate (Grade <3), severe (Grade 3), life-threatening (Grade 4), or fatal (Grade 5).
  Since the protocol restricted AE reporting to only those events which met National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0 grading criteria of Grade 3 (moderate) or higher, any infection not reported as an AE was assigned a severity of Grade <3 (effectively combining Grades 1 and 2); all other infections utilized the assigned CTCAE severity grade of the corresponding AE. A higher severity grade indicates a more severe event.
Time Frame: Up to 24 months post-transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 15 | 12
Participants
  Grade < 3 (Mild to Moderate) | 4 | 4
  Grade 3 (Severe) | 8 | 7
  Grade 4 (Life-threatening or Disabling) | 1 | 0
  Grade 5 (Fatal) | 2 | 1
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Test type: Superiority; p = 0.502, Cochran-Mantel-Haenszel

13. Secondary Outcome: Percent of Participants Experiencing a Serious Adverse Event (SAE) Related to Rituximab
Description: The percentage of participants with Serious Adverse Events (SAEs) as determined by the trial's medical monitor to be related to rituximab is reported.
Time Frame: Up to 35 months post-transplant
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percent of Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 15 | 12
Percent of Participants | 73.3 [54.6 to 92.1] | 58.3 [34.9 to 81.7]
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Test type: Superiority; p = 0.448, Fisher Exact

ADVERSE EVENTS:
Time Frame: Up to 35 months post-transplant
Description: Only adverse events grade 3 or higher were collected. Information was recorded by the site on the AE/SAE electronic Case Report Form (eCRF). All SAEs were to be reported within 24 hours of awareness, regardless of relationship to study procedures/therapy or expectedness of the event. SAEs included death, life-threatening events, hospitalization (or prolongation), inability to conduct normal life functions, birth defect, or condition requiring intervention to prevent these items.
Groups:
- Discontinued Pre-Transplant: Subjects who enrolled, but withdrew from the study prior to receiving a transplant.
- Discontinued Pre-Randomization: Subjects who were enrolled and transplanted on study, but withdrew from the study prior to randomization.
Arm/Group | Rituximab | Placebo | Discontinued Pre-Transplant | Discontinued Pre-Randomization
All-Cause Mortality (participants affected / at risk) | 2/15 | 3/12 | 4/11 | 2/7
Serious Adverse Events (participants affected / at risk) | 13/15 | 9/12 | 3/11 | 3/7
Other Adverse Events (participants affected / at risk) | 6/15 | 4/12 | 0/11 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=15) | Placebo (N=12) | Discontinued Pre-Transplant (N=11) | Discontinued Pre-Randomization (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Distal ileal obstruction syndrome (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transplant rejection (Immune system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocardiosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (5) | 4 (5) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Complications of transplant surgery (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thoracic cavity drainage (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=15) | Placebo (N=12) | Discontinued Pre-Transplant (N=11) | Discontinued Pre-Randomization (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sexually transmitted disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT02266888/Prot_001.pdf
  • Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT02266888/SAP_000.pdf